CLINICAL TRIAL: NCT00930943
Title: Effect of Extended-release Oxymorphone Hydrochloride (Opana® ER), Taken Fasting Versus With Food, on Cognitive Functioning in Opioid-tolerant Subjects: a Randomized, Single-blinded, Cross-over Study
Brief Title: Effect of Extended-release Oxymorphone Taken With or Without Food on Cognitive Functioning
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedVadis Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-133A
Record Dates: First submitted 2009-06-29; First posted 2009-07-02 (Estimated); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pain
Keywords: opioid tolerant; chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxymorphone ER 40 mg fed (Experimental): Participants received 40 mg oxymorphone ER after a high-fat meal of approximately 1,010 kCal
  Interventions: Drug: Oxymorphone ER
- Oxymorphone ER 40 mg fasting (Experimental): Participants received 40 mg oxymorphone ER after fasting for 8-12 hours
  Interventions: Drug: Oxymorphone ER

INTERVENTIONS:
Drug: Oxymorphone ER — 40 mg qd twice
  Other Names: Opana ER

SUMMARY:
The purpose of the study is to determine whether extended-release oxymorphone hydrochloride taken orally with a high-fat meal, generating an approximately 50% higher Cmax, impacts cognitive functioning, using Cambridge Neuropsychological Test Automated Battery (CANTAB) tests, to a greater extent than when taking under conditions of fasting.

DETAILED DESCRIPTION:
Oxymorphone 40 mg ER affects cognitive performance similarly within 3 hours post dose, whether given on an empty stomach or after a high-fat meal, suggesting that the altered pharmacokinetics, fed versus fasting and as described above, is not relevant for the medication's impact on cognition. Hence, the direction for oxymorphone ER to be dosed at least 1 hour before or 2 hours after eating, at least from a cognitive perspective, may be without merit.

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman, 18-65 years of age, inclusive
2. Able to provide informed consent and comply with all study procedures
3. Women of childbearing potential with a negative urine pregnancy test at screening and on adequate contraception
4. Chronic, non-malignant, painful condition, treated with long-acting opioid (methadone, OxyContin®, MS (Morphine Sulfate) Contin®, Kadian®, Avinza®, Fentanyl®, Opana® ER)
5. Opioid treatment for at least 3 months prior to screening at a minimum dose of 90 mg of morphine equivalents per day or 50 mcg of the fentanyl transdermal patch
6. Dose of opioid treatment stable for at least 1 week prior to screening and expected to be stable from screening through end of second testing
7. Weight at screening 100-300 pounds, inclusive

Exclusion Criteria:

1. Pregnant or breastfeeding
2. Gastrointestinal disorder or S/P gastrointestinal surgery impacting absorption of study medication (delayed gastric emptying, partial or complete gastrectomy)
3. Alcohol or substance abuse within 2 years of screening
4. Consumption of alcohol within 24 hours of a screening or testing visit
5. Consumption of xanthine-containing beverages (coffee, tea, coke) on the morning of a screening or testing visit
6. Impaired kidney or liver function (transaminase levels more than 3 times elevated; estimated creatinine clearance less than 50 mL/min)
7. Epworth sleepiness scale (ESS) score 16 or higher at screening
8. Medically concerning hypertension (≥ 160/100) or unstable cardiovascular illness
9. Any clinically significant illness that would interfere with study participation or put the subject at risk
10. Exposure to investigational medication within 30 days of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Egilius LH Spierings, MD, PhD, Principal Investigator — MedVadis Research Corporation
Locations (1):
- MedVadis Research Corporation, Wellesley Hills, Massachusetts, United States

REFERENCES:
- [Result] Spierings EL, Volkerts ER, Heitland I, Thomson H. A randomized, rater-blinded, crossover study of the effects of oxymorphone extended release, fed versus fasting, on cognitive performance as tested with CANTAB in opioid-tolerant subjects. Pain Med. 2014 Feb;15(2):264-71. doi: 10.1111/pme.12307. Epub 2013 Dec 11. PMID 24330343

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxymorphone 40 mg (Fed vs Fasting): After completion of the screening process and assuring eligibility in terms of inclusion/exclusion criteria, the subjects were randomized to determine at which testing visit a high-fat meal was to be consumed. (Note: randomization data are not available because old data records have been destroyed) They were instructed not to eat or drink, except for water, after midnight on the night before testing, not to consume alcohol within 24 hours of testing and xanthine-containing beverages (coffee, tea, coca cola, energy drinks, etc.) on the morning of the testing. Subjects who were taking an oral opioid were instructed not to take their morning dose on the days of testing, and those who used the transdermal fentanyl patch were instructed not to change the patch the night before.
  Each testing visit consisted of an assessment of adverse health and concomitant-medication changes and also a blood alcohol draw, followed by a high-fat breakfast, if applicable. Under supervision, the subjects took the study medication, a single dose of 40 mg oxymorphone ER, with water. Cognitive performance was assessed 1 hour and 3 hours post-dose using three Cambridge Neuropsychological Test Automated Battery (CANTAB) tests.
Period: Overall Study
Arm/Group | Oxymorphone 40 mg (Fed vs Fasting)
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Oxymorphone 40 mg (Fed vs Fasting): After completion of the screening process and assuring eligibility in terms of inclusion/exclusion criteria, the subjects were randomized to determine at which testing visit a high-fat meal was to be consumed. (Note: randomization data are not available) They were instructed not to eat or drink, except for water, after midnight on the night before testing, not to consume alcohol within 24 hours of testing and xanthine-containing beverages (coffee, tea, coca cola, energy drinks, etc.) on the morning of the testing. Subjects who were taking an oral opioid were instructed not to take their morning dose on the days of testing, and those who used the transdermal fentanyl patch were instructed not to change the patch the night before.
  Each testing visit consisted of an assessment of adverse health and concomitant-medication changes and also a blood alcohol draw, followed by a high-fat breakfast, if applicable. Under supervision, the subjects took the study medication, a single dose of 40 mg oxymorphone ER, with water. Cognitive performance was assessed 1 hour and 3 hours post-dose using three Cambridge Neuropsychological Test Automated Battery (CANTAB) tests.
Arm/Group | Oxymorphone 40 mg (Fed vs Fasting)
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
Pain Condition [Count of Participants; unit: Participants] — Number of Participants treated for the indicated condition. Participants may report more than one condition
  Participants
    Wrist pain | 1
    Flank pain | 1
    Chronic migraine | 2
    Neck pain | 4
    Low back pain | 21
    Leg pain | 5
    Fibromyalgia | 1
    Knee pain | 3
    Hip pain | 4
    Shoulder pain | 1
Opioid use [Count of Participants; unit: Participants] — Opioid used as treatment for chronic pain condition. Participants may take more than one opioid.
  Participants
    Oxycodone | 16
    Morphine | 4
    Meperidine | 1
    Methadone | 12
    Propoxyphene | 1
    Fentanyl | 5
    Codeine | 1
    Hydromorphone | 1
    Hydrocodone | 1
Opioid dose in morphine equivalent [Mean (Standard Deviation); unit: mg] | 206.8 (112.1)

OUTCOME MEASURES:

1. Primary Outcome: Rapid Visual Information Processing (RVP) Sensitivity [A']
Description: RVP is a test of sustained attention. It is a sensitive measure of general cognitive performance. A white box appears in the center of the computer screen, inside which digits, from 2 to 9, appear in a pseudorandom order, at the rate of 100 digits per minute. The subject is requested to detect target sequences of three digits (for example, 2-4-6, 3-5-7, 4-6-8) and to register responses using the response box. The two main outcome measures are the probability to detect the predefined sequence (sensitivity [A']) and the speed at which the sequence is registered (response latency [ms]).
Time Frame: 1 and 3 hours postdose
Population: Completers
Measure: Mean (Standard Error); unit: probability of detecting sequence
Groups:
- Oxymorphone 40 mg With High-fat Meal: Participants were instructed not to eat or drink, except for water, after midnight on the night before testing, not to consume alcohol within 24 hours of testing and xanthine-containing beverages (coffee, tea, coca cola, energy drinks, etc.) on the morning of the testing. Subjects who were taking an oral opioid were instructed not to take their morning dose on the days of testing, and those who used the transdermal fentanyl patch were instructed not to change the patch the night before.
  Each testing visit consisted of an assessment of adverse health and concomitant-medication changes and also a blood alcohol draw, followed by a high-fat breakfast. Under supervision, the subjects took the study medication, a single dose of 40 mg oxymorphone ER, with water. Cognitive performance was assessed 1 hour and 3 hours post-dose using three Cambridge Neuropsychological Test Automated Battery (CANTAB) tests.
- Oxymorphone 40 mg Fasting: Participants were instructed not to eat or drink, except for water, after midnight on the night before testing, not to consume alcohol within 24 hours of testing and xanthine-containing beverages (coffee, tea, coca cola, energy drinks, etc.) on the morning of the testing. Subjects who were taking an oral opioid were instructed not to take their morning dose on the days of testing, and those who used the transdermal fentanyl patch were instructed not to change the patch the night before.
  Each testing visit consisted of an assessment of adverse health and concomitant-medication changes and also a blood alcohol draw. Under supervision, the subjects took the study medication, a single dose of 40 mg oxymorphone ER, with water. Cognitive performance was assessed 1 hour and 3 hours post-dose using three Cambridge Neuropsychological Test Automated Battery (CANTAB) tests.
Arm/Group | Oxymorphone 40 mg With High-fat Meal | Oxymorphone 40 mg Fasting
Number analyzed (Participants) | 30 | 30
probability of detecting sequence
  1-hour post dose | 0.94 (0.01) | 0.93 (0.01)
  3-hours post dose | 0.95 (0.01) | 0.96 (0.01)
Statistical Analysis 1: Comparison: Oxymorphone 40 mg With High-fat Meal vs Oxymorphone 40 mg Fasting; The a priori sample-size estimation for a power of 80% with alpha = 0.05 was based on the primary-outcome measure, the rapid visual information processing (RVP) sensitivity (A') score. Using a repeated-measure ANOVA for the food effect (fed versus fasting) and assuming an effect size of f =0.26 generated a required sample size of 32 participants. However, only 30 subjects completed both testing visits, generating a power of 78.2%; Test type: Superiority; p < 0.001, ANOVA — repeated-measure ANOVA tested time-post-dose effect for Rapid Visual Information Processing (RVP): sensitivity (A'); (F[1,28] = 22.71; η2 = 0.45)
Statistical Analysis 2: Comparison: Oxymorphone 40 mg With High-fat Meal vs Oxymorphone 40 mg Fasting; Test type: Superiority; p = 0.01, ANOVA — repeated-measure ANOVA tested food x time-post-dose effect for Rapid Visual Information Processing (RVP): sensitivity (A'); F[1,28]=6.88; η2=0.20
Statistical Analysis 3: Comparison: Oxymorphone 40 mg With High-fat Meal vs Oxymorphone 40 mg Fasting; Test type: Superiority; p > 0.05, ANOVA — repeated-measure ANOVA testing food effect for Rapid Visual Information Processing (RVP): sensitivity (A')

2. Primary Outcome: Rapid Visual Information Processing (RVP) Response Latency
Description: as for outcome 1
Time Frame: 1 and 3 hours postdose
Population: Completers
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | Oxymorphone 40 mg With High-fat Meal | Oxymorphone 40 mg Fasting
Number analyzed (Participants) | 30 | 30
milliseconds
  1-hour post dose | 447.52 (17.47) | 455.96 (18.63)
  3-hours post dose | 422.33 (15.21) | 424.62 (18.84)
Statistical Analysis 1: Comparison: Oxymorphone 40 mg With High-fat Meal vs Oxymorphone 40 mg Fasting; Test type: Superiority; p < 0.001, ANOVA — Repeated-measure ANOVA testing time-post-dose effect for Rapid Visual Information Processing (RVP): response latency; (F[1,28] = 14.05; η2 = 0.33)
Statistical Analysis 2: Comparison: Oxymorphone 40 mg With High-fat Meal vs Oxymorphone 40 mg Fasting; Test type: Superiority; p > 0.05, ANOVA — repeated-measure ANOVA testing "food" and "food x time post dose" effect for Rapid Visual Information Processing (RVP): response latency

3. Secondary Outcome: Spatial Recognition Memory (SRM) Test Percentage of Correct Hits
Description: SRM tests visual spatial recognition memory in a two-choice forced discrimination paradigm. The subject is presented with a white square, which appears in sequence at five different locations on the screen. In the recognition phase, the subject sees a series of five pairs of squares, one of which is in a place previously seen in the presentation phase. The other square is in a location not seen in the presentation phase. Locations are tested in the reverse of the presentation order. The two main outcome measures are the percentage of correct trials (correct hits [%]) and the speed of the subject's response (response latency [ms]).
Time Frame: 1 and 3 hours postdose
Population: completers
Measure: Mean (Standard Error); unit: percentage of hits
Arm/Group | Oxymorphone 40 mg With High-fat Meal | Oxymorphone 40 mg Fasting
Number analyzed (Participants) | 30 | 30
percentage of hits
  1-hour post dose | 81.67 (1.78) | 83.17 (1.37)
  3-hours post dose | 80.50 (1.36) | 81.83 (1.94)
Statistical Analysis 1: Comparison: Oxymorphone 40 mg With High-fat Meal vs Oxymorphone 40 mg Fasting; Test type: Superiority; p > 0.05, ANOVA — repeated-measure ANOVA testing "food", "time-post-dose", and "food x time-post-dose" effect for SRM percentage of correct hits

4. Secondary Outcome: Spatial Recognition Memory (SRM) Test Response Latency
Description: as for outcome 3
Time Frame: 1 and 3 hours postdose
Population: completers
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | Oxymorphone 40 mg With High-fat Meal | Oxymorphone 40 mg Fasting
Number analyzed (Participants) | 30 | 30
milliseconds
  1-hour post dose | 1843.87 (98.05) | 1907.21 (104.05)
  3-hours post dose | 1555.51 (60.72) | 1606.26 (61.31)
Statistical Analysis 1: Comparison: Oxymorphone 40 mg With High-fat Meal vs Oxymorphone 40 mg Fasting; Test type: Superiority; p < 0.001, ANOVA — Repeated-measure ANOVA testing time-post-dose effect for Spatial Recognition Memory (SRM) response latency; (F[1,28] = 31.26; η2 = 0.53)
Statistical Analysis 2: Comparison: Oxymorphone 40 mg With High-fat Meal vs Oxymorphone 40 mg Fasting; Test type: Superiority; p > 0.05, ANOVA — repeated-measure ANOVA testing "food" and "food x time-post-dose" effect for SRM response latency

5. Secondary Outcome: Spatial Working Memory (SWM) Test Total Errors
Description: SWM is a test of the subject's ability to retain spatial information and to manipulate remembered items in working memory. It is a self-ordered task, which also assesses heuristic strategy. The test is a sensitive measure of executive function. It begins with a number of colored squares (boxes) being shown on the screen. By touching the boxes and using a process of elimination, the subject finds blue tokens in a number of boxes and uses them to fill up an empty column on the screen. The number of boxes is gradually increased, until it is necessary to search a total of eight boxes. The color and position of the boxes are changed from trial to trial to discourage the use of stereotyped search strategies. The two main outcome measures are errors (touching boxes that have been found to be empty and revisiting boxes that have already been found to contain a token - total errors) and a measure of strategy (strategy score).
Time Frame: 1 and 3 hours postdose
Population: completers
Measure: Mean (Standard Error); unit: number of errors
Arm/Group | Oxymorphone 40 mg With High-fat Meal | Oxymorphone 40 mg Fasting
Number analyzed (Participants) | 30 | 30
number of errors
  1-hour post dose | 40.00 (5.05) | 38.63 (4.45)
  3-hours post dose | 35.73 (4.70) | 37.40 (4.52)
Statistical Analysis 1: Comparison: Oxymorphone 40 mg With High-fat Meal vs Oxymorphone 40 mg Fasting; Test type: Superiority; p > 0.05, ANOVA — repeated-measure ANOVA testing "food", "time-post-dose", and "food x time-post-dose" effect for SWM total errors

6. Secondary Outcome: Spatial Working Memory (SWM) Test Strategy Score
Description: SWM is a test of the subject's ability to retain spatial information and to manipulate remembered items in working memory. The test is a sensitive measure of executive function. It begins with a number of colored squares (boxes) being shown on the screen. By touching the boxes and using a process of elimination, the subject finds blue tokens in a number of boxes and uses them to fill up an empty column on the screen. The number of boxes is gradually increased, until it is necessary to search a total of eight boxes. The color and position of the boxes are changed from trial to trial to discourage the use of stereotyped search strategies. The two main outcome measures are errors (touching boxes that have been found to be empty and revisiting boxes that have already been found to contain a token - total errors) and a measure of strategy (For assessed problems with six boxes or more, the number of distinct boxes used by the subject to begin a new search for a token)
Time Frame: 1 and 3 hours postdose
Population: completers
Measure: Mean (Standard Error); unit: number of boxes
Arm/Group | Oxymorphone 40 mg With High-fat Meal | Oxymorphone 40 mg Fasting
Number analyzed (Participants) | 30 | 30
number of boxes
  1-hour post dose | 35.13 (1.08) | 35.43 (1.04)
  3-hours post dose | 35.50 (1.16) | 35.57 (1.10)
Statistical Analysis 1: Comparison: Oxymorphone 40 mg With High-fat Meal vs Oxymorphone 40 mg Fasting; Test type: Superiority; p > 0.05, ANOVA — repeated-measure ANOVA testing "food", "time-post-dose", and "food x time-post-dose" effect for SWM strategy score

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Oxymorphone 40 mg With High-fat Meal | Oxymorphone 40 mg Fasting
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes